CLINICAL TRIAL: NCT02772094
Title: Autologous Dendritic Cell-Based Adjuvant Immunotherapy of Malignant Gliomas (WHO Grade IV Glioblastoma Multiforme) - Phase II Clinical Trial
Brief Title: Dendritic Cell-Based Tumor Vaccine Adjuvant Immunotherapy of Human Glioblastoma Multiforme (WHO Grade IV Gliomas)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Den-Mei Brain Tumor Education Foundation, Taichung, Taiwan (Unknown); Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Principal Investigator, Wen-Kuang Yang, MD PhD, Medical Chair Professor, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMR94-IRB-043-1
Record Dates: First submitted 2016-02-03; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Glioblastoma Multiforme; Glioblastoma
Keywords: glioblastoma multiforme; glioblastoma; newly diagnosed glioblastoma; immunotherapy; dendritic cells; grade IV astrocytoma; oncology; neurology; glioma; brain tumor; ADCTA-G
MeSH Terms: conditions — Glioblastoma; Neoplasms; Glioma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm, open-label (Experimental): Experimental:
  ADCTA-G total 10 doses, each dose (30+/-5 millions autologous dendritic cells plus 6+/-0.5 millions 100Gy-irradiated short-term cultured autologous GBM tumor cells) divided in 2 halves for subcutaneous injection into both axillar areas, in a course of 6 months (sequential series of weekly injections 4 times, bi-weekly injections twice; then monthly injections 4 times.
  Experimental: ADCTA-G total 10 doses, each dose (similar fore-mentioned numbers of 5:1 ratio of autologous dendritic cells and irradiated short-term cultured autologous GBM tumor cells) divided into 2 injections administered subcutaneously in both axillar areas, in a course of 8 months (sequential series of bi-weekly injections 4 times, then monthly injections 6 times).
  Interventions: Biological: Single arm, open-label

INTERVENTIONS:
Biological: Single arm, open-label — Biological: ADCTA-G. Biological: autologous DC loaded with irradiated autologous tumor cells. Biological: dendritic cell "vaccine". Drug: 180mg/m2•per day temozolomide prior and concomitant with radiotherapy. Radiotherapy: Local ionizing radiation 200 centigray(cGy)/day, 5 successive days per week for 6 weeks, total dose of 6000 cGy.
  Drug: Adjuvant chemotherapy-temozolomide (TMZ) monthly cycle, 200mg/m2•per day continued for 5 days in the beginning of every month, 6 cycles of TMZ.
  Other Names: ADCTA-G

SUMMARY:
Purposes:

The purpose of this phase-II clinical trial is to determine whether or not ADCTA-G, a biologic "vaccine" preparation of patient's own dendritic cell (DC) for glioblastoma multiforme (GBM) treatment, is safe and effective in extending the GBM patient's life. The current conventional multi-modal regimen that may include surgery for tumor resection or biopsy, temozolomide (TMZ) combined chemo-radiotherapy (CCRT) and TMZ adjuvant chemotherapy almost always leaves residual GBM cells to cause fatal recurrence, leading to medium survival period of 8 -15 months and over-all survival rates of about 30% in 2 years and <3% in 5 years after diagnosis/surgery. Thus, in neurosurgical oncology practice, GBM patients in the first 2-year period during and after receiving multi-modal therapy are watched closely for possible GBM tumor recurrence and mortal disease relapse and immediately given palliative treatments and health care, until death. In this phase-II trial, GBM patient participants who receive ADCTA-G "vaccine" adjuvant immunotherapy (added to the conventional multi-modal regimen) will be similarly watched closely by treatments and health care visits at least biweekly from the date of surgery/diagnosis to 24 months, and if alive followed by weekly phone calls and scheduled health care visits at least once every 3 months, up to 72 months after surgery. In the trial protocol, ADCT-G in 10 doses is administered after surgery, over a period of 6 or 8 months, as an adjuvant immunotherapy of the conventional multimodal regimen. Individual ADCTA-G "vaccine" lot of every participant GBM patient is manufactured from patient's own monocyte-derived dendritic cells and the patient's own tumor cell antigens, both of which are prepared by a distinct method of procedures performed within air particle-free barrier good laboratory practice (GLP) facility. Previous phase I/II clinical trial of ADCTA-G "vaccine" immunotherapy administered as an adjuvant to the conventional multimodal regimen, has obtained promising safety and efficacy results for GBM patients in a clinical center. This phase-II clinical trial in China Medical University Hospital-Taichung will employ essentially the same clinical protocols and the same distinct "vaccine" manufacturing method of standard operational procedures (SOP), that is, the conventional multimodal regimen plus adjuvant immunotherapy using personal ADCTA-G "vaccine" lot for every GBM patient participants.

DETAILED DESCRIPTION:
Rationale and Background :

Glioblastoma multiforme (GBM) and other WHO grade IV malignant gliomas of the brain are among the most lethal of human cancers. Despite current intensive multimodal regimen including the use of temozolomide (TMZ) for combined chemo-radiotherapy (CCRT) and for subsequent adjuvant chemotherapy, the medium survival period of GBM patients is still 8-16 months after diagnosis and surgery, with prognosis varied according to demographic features such as age, radiotherapy types and chemotherapy measures.These fatal brain cancers in general contain cancer cells with mutation in certain genes. Also, the mutated GBM cancer cells are usually heterogenous; and different GBM patients may have individual sets of heterogenous glioma cancer cells in which the mutant genes would generate altered antigens that can be recognized by the patient's adaptive immune system to mount immuno-targeting responses to reject or kill the GBM tumor cells. However, GBM is still fatal because it is highly immunosuppressive, i.e. able to anergize the immune effector cells in the body. Although surgical resection of rapidly expanding tumor bulk will prevent further physical damages to the brain and curtail the immunosuppression, the already anergized effector T lymphocytes still require functional restoration. On the other hand, post-surgical TMZ CCRT and adjuvant chemotherapy may weaken the residual tumor cells, but TMZ will also impair if not kill the active T lymphocytes in general, including anti-GBM lymphocytes. It is therefore important to exploit the adaptive immunity system for effective therapy of GBM. To apply the adaptive immunotherapy, it is best to use each patient's surgical tumor specimen to prepare the own individual "tumor regression antigens" for loading onto the patient's own dendritic cells (the "professional" antigen processing and presenting cells of the immune system). Dendritic cells loaded with tumor-specific antigens, upon maturation and inoculation ("vaccination"), would migrate/home to the T cell area of lymph nodes and stimulate proliferation of tumor-specific cytotoxic T lymphocyte that would move out of lymph node to find the brain tumor lesion to attack and eradicate the residual GBM tumor cells, resulting in prevention of GBM recurrence.

With fore-mentioned working hypotheses, the investigators carried out translational research from 1997 to 2002. A special method has been developed for production of an immunotherapeutic, which is named "autologous dendritic cell/autologous tumor cell antigens of GBM" (ADCTA-G). For clinical trial purpose, the investigators have established standard operational procedures (SOP) of the method with the use of clinical Good Manufacturing Practice (cGMP)-grade cytokines and pharmaceutical reagents. Individual ADCTA-G lots of all participant GBM patients are manufactured in high efficiency particle arresting (HEPA) air-filtered, germ-free bio-safety barrier clinical Good Laboratory Practice (cGLP) facilities. The phase I/II clinical trial was officially approved by Taiwan Department of Health and performed in a clinical center to demonstrate that ADCTA-G adjuvant immunotherapy was safe and apparently could prolong the survival for GBM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proved WHO grade-4 malignant glioma
2. Age: 13 years (physically mature) to 70 years
3. Karnofsky performance score before surgery: ≧70 [Karnofsky 1951] .
4. Adequate liver functions, including serum alanine aminotransferase (ALT or SGPT), serum aspartate aminotransferase (AST or SGOT), and alkaline phosphatase at ≤3.0 times upper limits of normal levels (ULN), total bilirubin ≤1.5mg/dl), total serum bilirubin <3 mg/dl
5. Adequate renal function (BUN ≤25 mg/ml; creatinine≤1.8 mg/dl，creatinine clearance >50 ml/min prior to starting therapy
6. Hemoblobin≧8 g/dl，platelet ≧100,000/μl，WBC>2,000/μl; absolute neutrophil count >1,000/μl
7. Prothrombin time and partial thromboplastin time≦1.5x the normal upper limit

Exclusion Criteria:

1. Pregnant or breast feeding
2. With radioactive implant
3. Acute infection, fever
4. Active collagen diseases
5. Acute cardiovascular diseases
6. Acute viral hepatitis
7. Syphilis
8. Human immunodeficiency virus (HIV) infection
9. Carrier of other transmissible infection
10. Immune deficiency due to chronic disease

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-05; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival with measures of medium survival period (in days) and annual survival rates (in %) | Post-recruitment surgery to death due to GBM or any other causes; close follow-up at leas by biweekly health care or emergency visits for 24 months, then weekly phone calls and scheduled visits at least every 3 months, up to 6 years after surgery
  The primary end-point is overall survival (OS), days measured from post-recruitment surgery date (tumor resection or biopsy) to date of death due to GBM or other causes, and if alive, to date of weekly phone calls and health care visit every 3 months, up to 6 years. Survival days of patients are depicted on Kaplan-Meier plots to show the medium survival period (days when 50% patients remained alive) and annual rates (% living patients per total) every year up to 5 years, and by log rank test to find statistical probability p value.
  Study groups of ADCTA-G immunotherapy plus conventional multimodal regimen will be compared to reference groups treated with conventional multimodal regimen (no ADCTA or other immunotherapy).
Adverse effects, acute and chronic, assessed according to NCI CTCAE Version 3 | Post-recruitment surgery to death, due to ADCTA-G, GBM disease or temozolomide chemotherapy; if alive, bi-weekly follow up for 24 months after surgery and then at least one visit in 3 months, up to 72 months
  Acute or delayed/chronic adverse effects, graded according to NCI CTCAE Version 3.0, e.g. temozolomide combined chemo-radiotherapy(CCRT)-/GBM-caused lymphopenia, measured by lymphocytes/microL blood, and by % of patients with lymphopenia of grade 1, 2, 3, or 4 severity.

SECONDARY OUTCOMES:
Disease progression-free period | From recruitment surgery to death, or if alive, biweekly for 24 months, and then weekly phone calls and at least once in 3 months, up to 72 months
  Progression-free survival period (days) is from date of surgery (tumor resection or biopsy) to date of neurological symptoms/signs relapse, verified by brain magnetic resonance (MRI) imaging, which is performed before and after surgery, and when symptoms and signs of disease progression occur, and subsequently one MRI scan in 3 months, till death or up to 6 years. The progression-free survival days of patient groups are depicted as Kaplan-Meier plots to show medium progression-free period (days when 50% patients remain free from GBM relapse) and annual rates (% progression-free patients of the total) from 1 to 5 years. Study groups of ADCTA-G immunotherapy plus conventional multimodal regimen will be compared to GBM reference groups with conventional therapy without immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Kuang Yang, M.D. PhD., Principal Investigator — China Medical University Hospital, Taichung Taiwan
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chang CN, Huang YC, Yang DM, Kikuta K, Wei KJ, Kubota T, Yang WK. A phase I/II clinical trial investigating the adverse and therapeutic effects of a postoperative autologous dendritic cell tumor vaccine in patients with malignant glioma. J Clin Neurosci. 2011 Aug;18(8):1048-54. doi: 10.1016/j.jocn.2010.11.034. Epub 2011 Jun 28. PMID 21715171